CLINICAL TRIAL: NCT06142487
Title: Prospective Double Blinded Randomized Assessment of the Effects of Silk Pillowcases on Acne Prone Skin
Brief Title: Assessment of the Effects of Silk Pillowcases on Acne Prone Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Responsible Party: Principal Investigator, Raja Sivamani, MD MS AP, Principle Investigator, Integrative Skin Science and Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: i23-11-silk_pillowcase_acne
Record Dates: First submitted 2023-11-13; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Acne Vulgaris
Keywords: acne; non-cystic acne; mild to moderate acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silk Pillowcase (Experimental): 100% Mulberry Silk Pillowcase used every night
  Interventions: Other: Silk Pillowcase
- Cotton Pillowcase (Active Comparator): 100% Cotton Pillowcase used every night
  Interventions: Other: Cotton Pillowcase

INTERVENTIONS:
Other: Silk Pillowcase — 100% Mulberry Silk Pillowcase
  Arms: Silk Pillowcase
Other: Cotton Pillowcase — 100% Cotton Pillowcase
  Arms: Cotton Pillowcase

SUMMARY:
The purpose of this study is to determine the effects of using silk pillowcases in mild to moderate non-cystic acne prone skin in comparison to cotton pillowcases.

DETAILED DESCRIPTION:
The investigators will evaluate acne severity/ lesion count, trans-epidermal water loss, and sebum production in participants. There is an equal chance of being assigned a 100% silk pillowcase or 100% cotton pillowcase.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 15-45 years of age
* The presence of mild to moderate acne vulgaris based on investigator global assessment
* Presence of at least 5 inflammatory lesions and at least 5 non-inflammatory lesions

Exclusion Criteria:

* The presence of severe acne as noted by investigator global assessment.
* Those who are unwilling to discontinue systemic antibiotics and benzoyl peroxide for 4 weeks meet the washout criteria prior to enrolling.
* Those who are unwilling to keep their facial regimen consistent throughout the study, and for 1 month prior to enrolling.
* Individuals who are unwilling to wash pillowcase every week using provided detergent.
* Use of isotretinoin within the three months prior to enrolment
* Individuals who primarily sleep on their back
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack year
* Individuals on oral contraceptive pills or progesterone or estrogen containing therapies.
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study
* Individuals with known allergy or sensitivity to Mulberry Silk or Cotton Fibers in fabric

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Acne Lesion Counts: Inflammatory Lesions | 8 weeks
  The inflammatory lesion counts will be counted and compared against baseline
Acne Lesion Counts: Non-Inflammatory Lesions | 8 weeks
  The non-inflammatory lesion counts will be counted and compared against baseline
Facial Erythema Intensity Score | 8 Weeks
  Facial erythema will be measured as the erythema intensity score as measured by the image analysis system (BTBP 3D Pro)

SECONDARY OUTCOMES:
Transepidermal water loss | 8 Weeks
  Change in Facial Trans-epidermal Water Loss, measured with vapometer
Sebum Excretion Rate | 8 weeks
  Shift in the facial sebum excretion rate, measured with sebumeter
Skin Microbiome, relative abundance of C. acnes | 8 Weeks
  Changes in skin microbiome relative abundance of C. acnes will be assessed with swab based collections of the facial skin microbiome
Skin Hydration | 8 Weeks
  Skin Hydration measured with MoistureMeter

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD MS AP, Principal Investigator — Study Principal Investigator

IPD SHARING:
Plan to Share IPD: No